CLINICAL TRIAL: NCT00873899
Title: Evolution of Management Strategies of Heart Failure Patients With Implantable Defibrillators
Acronym: EVOLVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regione Lombardia (Other)
Collaborators: CEFRIEL, Milan Italy (Unknown); Politecnico di Milano (Other); Medtronic Italia (Industry)
Responsible Party: Maurizio Marzegalli - Direttore Dipartimento DEA e UO Cardiologia, Azienda Ospedaliera San Carlo Borromeo
Other Study IDs: RFPS-2006-2-335243-UO RL
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Heart Failure; Sudden Cardiac Death; Implantable Defibrillator
Keywords: Heart Failure; Implantable defibrillator; Remote Monitoring
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Remote Arm: The patients in Remote arm will receive a Medtronic CareLink Monitor to perform remote interrogation and transmission of ICD data. The remote arm ICD will be programmed to transmit over the CareLink Network.
  Interventions: Device: The Medtronic CareLink system (Minneapolis, MN, USA).
- Implantable defibrillator patients: Heart failure patients implanted with a wireless-transmission-enabled ICD.
  Interventions: Device: The Medtronic CareLink system (Minneapolis, MN, USA).

INTERVENTIONS:
Device: The Medtronic CareLink system (Minneapolis, MN, USA). — The Medtronic CareLink system(Minneapolis, MN, USA)includes a patient monitor plugged into a standard analog telephone connection, and a lightweight wand to communicate with the implanted device. Interrogation of the device and transmission of the data occur when the patient places the wand over the implanted device. The system uses radio frequency telemetry for wireless automatic communication. This allows for data transmission without patient intervention and enables automatic transmissions at pre-specified routine intervals as well as alert-based downloads.The system can transmit data in case of programmable conditions on diagnostic variables, arrhythmias, delivered ICD therapies, battery/lead issues, and alert the physician via phone or e-mail. The patient's information is sent to a secure Network server via the telephone connection and clinical staff can review device information.Available data are equivalent to that which can be retrieved at an in-office visit.

SUMMARY:
The EVOLVO study is designed to compare the remote defibrillator management to the current standard of care, to assess its ability to treat and triage patients more effectively.

DETAILED DESCRIPTION:
Heart failure patients with implantable defibrillators (ICD) perform frequent clinic visits for routine device monitoring. Moreover, in case of clinical events, such as ICD shocks or alert notifications for changes in cardiac status or safety issues, they often visit the emergency department or the clinic for an unscheduled visit. These planned and unplanned visits create a great burden on healthcare providers. Internet-based remote device interrogation systems, allowing physician's remote access to patients' data, are being proposed for reducing routine and interim visits and for earlier detection and notification of alert conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with left ventricular systolic dysfunction, left ventricular ejection fraction ≤35%, as documented at the moment of ICD implant;
* Patient implanted with a wireless-transmission-enabled Medtronic ICD or CRT-D;
* Patient must be able and willing to replace regularly-scheduled in-office routine follow-ups with remote follow-ups;
* Patient must be able to attend all required follow-up visits at the study center.

Exclusion Criteria:

* Patient is less than 18 years of age;
* Patient is unwilling or unable to sign an informed consent;
* Patient life expectancy is less than 12 months;
* Patient is participating in another clinical study that may have an impact on the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with left ventricular systolic dysfunction implanted wih ICD
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
The rate of cardiac or device related clinic visits | 16 months

SECONDARY OUTCOMES:
Rate of visits related or not to episodes of worsening of heart failure. Rate and related costs of total health care utilizations (all planned and unplanned hospital admissions involving and not an overnight stay) for cardiac or device related events | one year

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Azienda Ospedaliera Spedali Civili, Brescia
  - Azienda Ospedaliera Niguarda Ca' Granda, Milan
  - Azienda Ospedaliera San Carlo Borromeo, Milan
  - IRCCS Auxologico Italiano Ospedale S. Luca, Milan
  - IRCCS San Raffaele, Milan
  - IRCCS Policlinico San Matteo, Pavia

REFERENCES:
- [Derived] Zanaboni P, Landolina M, Marzegalli M, Lunati M, Perego GB, Guenzati G, Curnis A, Valsecchi S, Borghetti F, Borghi G, Masella C. Cost-utility analysis of the EVOLVO study on remote monitoring for heart failure patients with implantable defibrillators: randomized controlled trial. J Med Internet Res. 2013 May 30;15(5):e106. doi: 10.2196/jmir.2587. PMID 23722666
- [Derived] Landolina M, Perego GB, Lunati M, Curnis A, Guenzati G, Vicentini A, Parati G, Borghi G, Zanaboni P, Valsecchi S, Marzegalli M. Remote monitoring reduces healthcare use and improves quality of care in heart failure patients with implantable defibrillators: the evolution of management strategies of heart failure patients with implantable defibrillators (EVOLVO) study. Circulation. 2012 Jun 19;125(24):2985-92. doi: 10.1161/CIRCULATIONAHA.111.088971. Epub 2012 May 24. PMID 22626743
- [Derived] Marzegalli M, Landolina M, Lunati M, Perego GB, Pappone A, Guenzati G, Campana C, Frigerio M, Parati G, Curnis A, Colangelo I, Valsecchi S. Design of the evolution of management strategies of heart failure patients with implantable defibrillators (EVOLVO) study to assess the ability of remote monitoring to treat and triage patients more effectively. Trials. 2009 Jun 18;10:42. doi: 10.1186/1745-6215-10-42. PMID 19538734